CLINICAL TRIAL: NCT00915304
Title: Patient Specific Automatic Reminders in Primary Care - the EBMeDS Randomised Trial
Brief Title: Evidence-Based Medicine Electronic Decision Support Study
Acronym: EBMeDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: The Finnish Medical Society Duodecim (Unknown); Finnish Institute for Health and Welfare (Other Government); Duodecim Medical Publications Ltd. (Industry); ProWellness Ltd. (Unknown); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Principal Investigator, Tiina Kortteisto, researcher, Tampere University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: EBMeDS-40344-06
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Decision Support Systems, Clinical
Keywords: Clinical Decision Support System; Automatic reminder; Primary care; Evidence-Based Medicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: The EBMeDS reminders — Phase I: EBMeDS reminders specific to the visiting or caring patient and his/her clinical problem are generated when the practitioner uses the electronic patient record. During visits of intervention group patients the EBMeDS reminders will be shown on screen to the practitioner.
  Phase II: As phase I and in addition, results of the Virtual Health Check (VHC) of all the intervention group patients will be shown to the practitioners.Phase II will be fulfilled in Autumn 2010 and follow-up time will be about 3 months.

SUMMARY:
The purpose of this study is to analyze the effect of the Evidence-Based Medicine electronic Decision Support (EBMeDS) automatic reminders in primary health care.

Hypothesis (1)is that in the intervention group the total number of EBMeDS reminders will decrease compared to the control group.

Hypothesis (2) is that in the intervention group the quality measures will increase faster compared to the control group at follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* All residents of Sipoo who have patient ID number in the Mediatri electronic patient record system in Sipoo Health Centre

Exclusion Criteria:

* Those residents who's occupational health care is produced by Sipoo Health Centre

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12101 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The number of reminders triggered (in relation to the number of eligible patients, Ri/Ni) during repeated Virtual Health Checks (VHCs) | Follow-up time max one and half year
  VHC will be performed once a week for the whole study population, beginning at baseline and before randomisation. The main outcome measure is Ri/Ni at follow-up time after commencement of the study where Ri is the total number of reminders triggered by the patient record data in intervention and in control group at the time of analysis, and Ni is the total number of patients.

SECONDARY OUTCOMES:
Specific clinical measures compared to an intervention and a control group
  Clinical measures as mean values of laboratory parameters, for example a mean level of HbA1c, a mean level of total cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Rissanen, Professor, Study Director — University of Tampere; School of Health Sciences; Tiina Kortteisto, MSc, Principal Investigator — University of Tampere; School of Health Sciences
Locations (1):
- University of Tampere; School of Health Sciences, Tampere, Finland, Finland

REFERENCES:
- [Derived] Kortteisto T, Raitanen J, Komulainen J, Kunnamo I, Makela M, Rissanen P, Kaila M; EBMeDS (Evidence-Based Medicine electronic Decision Support) Study Group. Patient-specific computer-based decision support in primary healthcare--a randomized trial. Implement Sci. 2014 Jan 20;9:15. doi: 10.1186/1748-5908-9-15. PMID 24444113
- See also: Click here for more information about this study and EDMeDS — http://www.ebmeds.org